CLINICAL TRIAL: NCT00015015
Title: Dichloroacetate Kinetics, Metabolism and Toxicology
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 7355-CP-001
Record Dates: First submitted 2001-04-17; First posted 2001-04-19 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Lactic Acidosis
Keywords: Dichloroacetate; Chlorinated hydrocarbons; Genetic disease; Toxicology; Biotransformation
MeSH Terms: conditions — Acidosis, Lactic; Genetic Diseases, Inborn | interventions — Dichloroacetic Acid

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Dichloroacetate

SUMMARY:
Dichloroacetate (DCA) is a product of water chlorination and a metabolite of certain industrial solvents, thus making it a chemical of environmental concern. However, DCA is also used as an investigational drug for treating various diseases of adults and children, at doses far greater than those to which humans are normally exposed in the environment. Our research involves how DCA is metabolized by healthy adults and by children with a fatal genetic disease, congenital lactic acidosis (CLA) who are treated with DCA.

ELIGIBILITY:
Children with congenital lactic acidosis Healthy adult volunteers

Ages: 3 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1994-12; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (1):
- Univ. of Florida, Gainesville, Florida, United States